CLINICAL TRIAL: NCT02437968
Title: Disseminating Evidence-based Practice to the Schools: CBT for Child Anxiety
Acronym: Cats&Dogs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH086438
Record Dates: First submitted 2015-04-20; First posted 2015-05-08 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wave 1 (Experimental): South New Jersey school service providers.
  Interventions: Behavioral: Camp Cope-A-Lot (Computer-assisted CBT program)
- Wave 2 (Experimental): Philadelphia suburbs and surrounding community service providers
  Interventions: Behavioral: Camp Cope-A-Lot (Computer-assisted CBT program)
- Wave 3 (Experimental): Mississauga, ON (Canada) school district service providers.
  Interventions: Behavioral: Camp Cope-A-Lot (Computer-assisted CBT program)

INTERVENTIONS:
Behavioral: Camp Cope-A-Lot (Computer-assisted CBT program) — Camp Cope-A-Lot is a computer-assisted program that includes psychoeducation and clinician guided exposure tasks for anxious children.

SUMMARY:
The present study aims to test the implementation and sustainability of (a) a Computer-Assisted Cognitive-Behavioral Treatment (CACBT) for youth anxiety and (b) the BASC-2 TRS to identify anxious youth in the school setting using a cohort-sequential design (i.e., three years at 20 schools over the span of five years).

'Camp Cope-A-Lot (Computer-assisted CBT program)'

DETAILED DESCRIPTION:
The present study will test the implementation and sustainability of (a) a Computer-Assisted Cognitive-Behavioral Treatment (CACBT) for youth anxiety and (b) the BASC-2 TRS to identify anxious youth in the school setting using a cohort-sequential design (i.e., three years at 20 schools over the span of five years). There are 3 phases: Phase I (baseline): Gather data on prevalence and services provided via screening measures and treatment trackers: Phase II (implementation): Train school staff in the identification of anxious youth (i.e. BASC-2 TRS) and the provision of the intervention (i.e., CACBT), modifying assessment and treatment procedures so as to best fit each individual school. Identify barriers and facilitators of implementation by gathering the qualitative experience of school staff: Phase II (sustainability): Discontinue training and supervision. Assess sustainability of the assessment and intervention. Identify barriers and facilitators of implementation by gathering the qualitative experience of school staff.

'Camp Cope-A-Lot (Computer-assisted CBT program)"

ELIGIBILITY:
Inclusion Criteria:

* All mental health workers (e.g., guidance, social work, school psychologists) in the schools will be eligible to be trained.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in the number of children identified as anxious. | Baseline, end of year 1, end of year 2, end of year 3
Change in the number of children treated for anxiety. | Baseline, end of year 1, end of year 2, end of year 3